CLINICAL TRIAL: NCT00219128
Title: An Eight-week, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter Study Comparing Aliskiren 150 mg, 300 mg, and 600 mg to Placebo in Patients With Essential Hypertension
Brief Title: A Dose Ranging Study to Compare the Safety and Efficacy of Aliskiren 150mg, 300mg, and 600mg to Placebo in Patients With High Blood Pressure.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2308
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, placebo
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
Evaluate the blood pressure lowering effect of aliskiren 150mg, 300mg and 600mg compared to placebo in patients with essential hypertension

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients who are eligible and able to participate in the study

Exclusion Criteria

* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident.

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2004-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 8 weeks
Diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 4 weeks and 8 weeks
Blood pressure <140/90 mmHg after 4 weeks and 8 weeks
Evaluate potential return of hypertension at 4 days and 2 weeks after 8 weeks
Evaluate high and low level drug effect using 24 hour blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States